CLINICAL TRIAL: NCT06154083
Title: The Impact of Ovarian Stimulation Intensity on Embryo Euploidy in Advanced Age Women
Brief Title: INtensity of OVarian Stimualtion and Euploid Embryos
Acronym: INOVEE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-INO-2023-14; 2023-507028-22 (EudraCT Number)
Record Dates: First submitted 2023-11-13; First posted 2023-12-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Fertility
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follitropin-delta 20 mcg/day from D1 (Experimental)
  Interventions: Drug: Follitropin-delta (Rekovelle) 20 mcg/day from D1
- Follitropin-delta 15 mcg/day from D1 (Active Comparator)
  Interventions: Drug: Follitropin-delta (Rekovelle) 15 mcg/day from D1

INTERVENTIONS:
Drug: Follitropin-delta (Rekovelle) 20 mcg/day from D1 — On day 2 or 3 of the menstrual cycle, daily injections of 20 mcg of Rekovelle (Stimulation Day 1) will be administered. Scan controls blood exams are performed on stimulation days 6, 8, 10 and, according to clinical needs, until trigger day. The dose will be the same during the whole course of stimulation and no dose adjustments will be performed.
  Arms: Follitropin-delta 20 mcg/day from D1
Drug: Follitropin-delta (Rekovelle) 15 mcg/day from D1 — On day 2 or 3 of the menstrual cycle, daily injections of 15 mcg of Rekovelle (Stimulation Day 1) will be administered. Scan controls and blood exams are performed on stimulation days 6, 8, 10 and, according to clinical needs, until trigger day. The dose will be the same during the whole course of stimulation and no dose adjustments will be performed.
  Arms: Follitropin-delta 15 mcg/day from D1

SUMMARY:
This randomized trial was designed as a no-inferiority trial aiming to evaluate if the intensity of stimulation (a milder vs a more intense approach) may have an impact on the number of euploid embryos and the morpho kinetic parameters in advanced age women undergoing PGT-A with a PPOS protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients with indication for IVF
* Undergoing preimplantation genetic screening cycles
* AMH >= 1.5 ng/ml and < 3.5 ng/ml (AMH result of up to one year will be valid)
* BMI 18.5 - 30 Kg/m2

Exclusion Criteria:

* Severe male factor requiring TESE (testicular sperm extraction)
* AMH < 1.5 ng/ml or >= 3.5 ng/ml
* Administration of any other drug potentially interfering with the treatment
* Contraindication for hormonal treatment
* Recent history of severe disease requiring regular treatment (clinically significant concurrent medical condition that could compromise subject safety or interfered with the trial assessment).
* Monogenic disease to be detected with PGT-M

Ages: 38 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Number of euploid embryos | Trough study completion, an average of 20-30 days.
  Number of euploid embryos

SECONDARY OUTCOMES:
Gonadotropin dose | Up to oocyte pickup, an average of 10-20 days
  Total gonadotropin dose used
Length of stimulation | Up to oocyte pickup, an average of 10-20 days
  Days of stimulation
Estradiol | Up to oocyte pickup, an average of 10-20 days
  Estradiol level
Progesterone | Up to oocyte pickup, an average of 10-20 days
  Progesterone level
LH | Up to oocyte pickup, an average of 10-20 days
  LH level
Follicular Output RaTe (FORT) | Day one of stimulation. 1 Day
  ratio of the number of preovulatory follicles and the number of antral follicles available at the start of stimulation
Cycle cancelation rate | Up to oocyte pickup, an average of 10-20 days
  Cycle cancelation rate
Fertilization rate | Up to one day after oocyte pickup, an average of 10-20 days
  Fertilization rate
Time of appearance of the 2nd polar body (tPB2) | Up to one day after oocyte pickup, an average of 10-20 days
  Time of appearance of the 2nd polar body (tPB2)
Time of pronuclei disappearance (tPNf) | Up to one day after oocyte pickup, an average of 10-20 days
Time of division from 2 to 8 cells | Until 1, or 4 days after insemination
Time of compactation (tSC) | Until 3, or 4 days after insemination
Time of morula (tM) | Until 4 or 7 days after insemination
Time of cavitation (tSB) | Until 4 or 7 days after insemination
Time of full blastulation (tB) | Until 4 or 7 days after insemination
Total number of day 5 blastocysts | Until 5, 6 or 7 days after insemination
Total number of good quality blastocysts | Until 5, 6 or 7 days after insemination
Total number of embryos | Until 5, 6 or 7 days after insemination
Blastocyst formation rate | Until 5, 6 or 7 days after insemination
  proportion of 2PN zygotes that reach the blastocyst stage
Number of embryos cryopreserved | Until 5, 6 or 7 days after insemination
Embryo stage | Until 5, 6 or 7 days after insemination
Clinical pregnancy rate | 5-6 weeks after transfer
  defined as the visualization of one or more gestational sacs
Ongoing pregnancy rate | 8-10 weeks after transfer
  defined as a viable intrauterine pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alper MM, Fauser BC. Ovarian stimulation protocols for IVF: is more better than less? Reprod Biomed Online. 2017 Apr;34(4):345-353. doi: 10.1016/j.rbmo.2017.01.010. Epub 2017 Jan 24. PMID 28169189
- [Background] Arce JC, Larsson P, Garcia-Velasco JA. Establishing the follitropin delta dose that provides a comparable ovarian response to 150 IU/day follitropin alfa. Reprod Biomed Online. 2020 Oct;41(4):616-622. doi: 10.1016/j.rbmo.2020.07.006. Epub 2020 Jul 15. PMID 32819842
- [Background] Baart EB, Martini E, Eijkemans MJ, Van Opstal D, Beckers NG, Verhoeff A, Macklon NS, Fauser BC. Milder ovarian stimulation for in-vitro fertilization reduces aneuploidy in the human preimplantation embryo: a randomized controlled trial. Hum Reprod. 2007 Apr;22(4):980-8. doi: 10.1093/humrep/del484. Epub 2007 Jan 4. PMID 17204525
- [Background] Briggs R, Kovacs G, MacLachlan V, Motteram C, Baker HW. Can you ever collect too many oocytes? Hum Reprod. 2015 Jan;30(1):81-7. doi: 10.1093/humrep/deu272. Epub 2014 Oct 31. PMID 25362088
- [Background] Devesa M, Tur R, Rodriguez I, Coroleu B, Martinez F, Polyzos NP. Cumulative live birth rates and number of oocytes retrieved in women of advanced age. A single centre analysis including 4500 women >/=38 years old. Hum Reprod. 2018 Nov 1;33(11):2010-2017. doi: 10.1093/humrep/dey295. PMID 30272168
- [Background] Franasiak JM, Forman EJ, Hong KH, Werner MD, Upham KM, Treff NR, Scott RT Jr. The nature of aneuploidy with increasing age of the female partner: a review of 15,169 consecutive trophectoderm biopsies evaluated with comprehensive chromosomal screening. Fertil Steril. 2014 Mar;101(3):656-663.e1. doi: 10.1016/j.fertnstert.2013.11.004. Epub 2013 Dec 17. PMID 24355045
- [Background] Irani M, Canon C, Robles A, Maddy B, Gunnala V, Qin X, Zhang C, Xu K, Rosenwaks Z. No effect of ovarian stimulation and oocyte yield on euploidy and live birth rates: an analysis of 12 298 trophectoderm biopsies. Hum Reprod. 2020 May 1;35(5):1082-1089. doi: 10.1093/humrep/deaa028. PMID 32348476
- [Background] Kok JD, Looman CW, Weima SM, te Velde ER. A high number of oocytes obtained after ovarian hyperstimulation for in vitro fertilization or intracytoplasmic sperm injection is not associated with decreased pregnancy outcome. Fertil Steril. 2006 Apr;85(4):918-24. doi: 10.1016/j.fertnstert.2005.09.035. PMID 16580375
- [Background] La Marca A, Minasi MG, Sighinolfi G, Greco P, Argento C, Grisendi V, Fiorentino F, Greco E. Female age, serum antimullerian hormone level, and number of oocytes affect the rate and number of euploid blastocysts in in vitro fertilization/intracytoplasmic sperm injection cycles. Fertil Steril. 2017 Nov;108(5):777-783.e2. doi: 10.1016/j.fertnstert.2017.08.029. Epub 2017 Oct 4. PMID 28987789
- [Background] Neves AR, Montoya-Botero P, Sachs-Guedj N, Polyzos NP. Association between the number of oocytes and cumulative live birth rate: A systematic review. Best Pract Res Clin Obstet Gynaecol. 2023 Mar;87:102307. doi: 10.1016/j.bpobgyn.2022.102307. Epub 2022 Dec 27. PMID 36707342
- [Background] Polyzos NP, Drakopoulos P, Parra J, Pellicer A, Santos-Ribeiro S, Tournaye H, Bosch E, Garcia-Velasco J. Cumulative live birth rates according to the number of oocytes retrieved after the first ovarian stimulation for in vitro fertilization/intracytoplasmic sperm injection: a multicenter multinational analysis including approximately 15,000 women. Fertil Steril. 2018 Sep;110(4):661-670.e1. doi: 10.1016/j.fertnstert.2018.04.039. PMID 30196963
- [Background] Ubaldi FM, Cimadomo D, Vaiarelli A, Fabozzi G, Venturella R, Maggiulli R, Mazzilli R, Ferrero S, Palagiano A, Rienzi L. Advanced Maternal Age in IVF: Still a Challenge? The Present and the Future of Its Treatment. Front Endocrinol (Lausanne). 2019 Feb 20;10:94. doi: 10.3389/fendo.2019.00094. eCollection 2019. PMID 30842755
- [Background] Venetis CA, Tilia L, Panlilio E, Kan A. Is more better? A higher oocyte yield is independently associated with more day-3 euploid embryos after ICSI. Hum Reprod. 2019 Jan 1;34(1):79-83. doi: 10.1093/humrep/dey342. PMID 30476100
- [Background] Wu Q, Li H, Zhu Y, Jiang W, Lu J, Wei D, Yan J, Chen ZJ. Dosage of exogenous gonadotropins is not associated with blastocyst aneuploidy or live-birth rates in PGS cycles in Chinese women. Hum Reprod. 2018 Oct 1;33(10):1875-1882. doi: 10.1093/humrep/dey270. PMID 30137360
- See also: Related Info — http://www.dexeus.com